CLINICAL TRIAL: NCT06668961
Title: A Phase II Clinical Study to Evaluate the Safety and Efficacy of SI-B001+SI-B003 Combined With Platinum-based Chemotherapy (SI-B001+SI-B003+ Platinum-based Chemotherapy) as First-line Treatment in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of SI-B001+SI-B003 Combined With Platinum-based Chemotherapy as First-line Treatment in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001-SI-B003-203
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Participants will receive treatment during the first cycle. Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: SI-B001; Drug: SI-B003
- Cohort B (Experimental): Participants will receive treatment during the first cycle. Participants with clinical benefit could receive additional treatment for more cycles. The administration will be terminated because of disease progression or intolerable toxicity occurring or other reasons.
  Interventions: Drug: SI-B001

INTERVENTIONS:
Drug: SI-B001 — Administration by intravenous infusion
Drug: SI-B003 — Administration by intravenous infusion
  Arms: Cohort A

SUMMARY:
This study is a open, multi-center phase II clinical study to explore the efficacy, safety and pharmacokinetic/pharmacodynamic characteristics of SI-B001+SI-B003 combined with platinum-based chemotherapy as first-line treatment in patients with recurrent or metastatic head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. Patients with recurrent or metastatic head and neck squamous cell carcinoma;
6. Consent to provide tumor tissue samples or fresh tissue samples archived from the primary or metastatic lesions within 2 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. Physical status score: ECOG ≤1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. No blood transfusion or colony-stimulating factor was allowed within 14 days before the first use of the study drug, and the organ function level must meet the requirements;
12. Coagulation function: international normalized ratio (INR) ≤1.5, and activated partial thromboplastin time (APTT) ≤1.5×ULN;
13. Urinary protein ≤1+ or ≤1000mg/24h;
14. Fertile female subjects, or male subjects with fertile partners, must use highly effective contraception from 7 days before the first dose until 24 weeks after the dose. Female subjects of childbearing potential had to have a negative serum pregnancy test within 7 days before the first dose.

Exclusion Criteria:

1. Squamous cell carcinoma of the nasopharynx, salivary gland, paranasal sinus, skin or of unknown primary site;
2. Patients with any of the following conditions were not eligible for the study: a) suitable and willing for local treatment; b) received systemic therapy, excluding treatment for locally advanced disease as part of multimodal therapy;
3. Patients with active central nervous system metastasis;
4. Who had participated in any other clinical trial within 4 weeks before the study dose;
5. Received radiotherapy within 4 weeks before the first dose of study drug;
6. Use of traditional Chinese medicine with anti-tumor indications within 2 weeks;
7. Had undergone major surgery within 4 weeks before the first dose;
8. Systemic corticosteroids or immunosuppressive agents were required within 2 weeks before study dosing;
9. Pulmonary disease was defined as ≥ grade 3 according to NCI-CTCAE v5.0; Patients with existing or a history of interstitial lung disease (ILD);
10. Have active infection requiring intravenous anti-infective therapy;
11. Had received immunotherapy and had grade ≥3 irAE or grade ≥2 immune-related myocarditis;
12. Received live attenuated vaccine within 4 weeks before the first dose of study drug;
13. Had taken an immunomodulatory drug within 14 days before the first dose of study drug;
14. Patients at risk for active autoimmune disease or with a history of autoimmune disease;
15. Other malignant tumors within 5 years before the first administration;
16. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
17. Poorly controlled hypertension;
18. Patients with poor blood glucose control before the first dose;
19. Had a history of severe cardiovascular and cerebrovascular diseases;
20. Previous history of allogeneic stem cell, bone marrow or organ transplantation;
21. Patients with massive or symptomatic effusions or poorly controlled effusions;
22. Patients with a history of allergy to recombinant humanized antibodies or to any of the excipients of SI-B001 or SI-B003;
23. Had severe infusion reactions to antibody therapy in the past;
24. Had autologous or allogeneic stem cell transplantation;
25. Pregnant or lactating women;
26. The investigator did not consider it appropriate to apply other criteria for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the participant's first dose of SI-B001+SI-B003 to the first date of either disease progression or death, whichever occurs first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally emerging, or any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition during the treatment of SI-B001+SI-B003. The type, frequency and severity of TEAE will be evaluated during the treatment of SI-B001+SI-B003.
Cmax | Up to approximately 24 months
  Maximum serum concentration (Cmax) of SI-B001+SI-B003 will be investigated.
Tmax | Up to approximately 24 months
  Time to maximum serum concentration (Tmax) of SI-B001+SI-B003 will be investigated.
Ctrough | Up to approximately 24 months
  Ctrough is defined as the lowest serum concentration of SI-B001+SI-B003 prior to the next dose will be administered.
Anti-drug antibody (ADA) | Up to approximately 24 months
  Frequency and titer of anti-SI-B001 and SI-B003 antibody (ADA) will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China